CLINICAL TRIAL: NCT02575794
Title: Phase 1 Dose Escalation and Drug Distribution Study of Oral Terameprocol in Patients With Recurrent High Grade Glioma
Brief Title: Terameprocol in Treating Patients With Recurrent High Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Erimos Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABTC-1401; IRB00065527 (Other: JHM IRB); UM1CA137443 (NIH)
Record Dates: First submitted 2015-10-09; First posted 2015-10-15 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: High Grade Glioma (III or IV)
MeSH Terms: conditions — Glioma | interventions — terameprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (terameprocol) (Experimental): Patients receive terameprocol PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study
  Interventions: Drug: Terameprocol; Other: Pharmacological Study

INTERVENTIONS:
Drug: Terameprocol — Given PO
  Other Names: 1,1'-(2,3-Dimethyl-1,4-butanediyl)bis(3,4-dimethoxybenzene); EM-1421; M4N; tetra-O-methyl NDGA; Tetra-O-methyl Nordihydroguaiaretic Acid; TMNDGA
Other: Pharmacological Study — Correlative studies
  Other Names: Pharnacological Study

SUMMARY:
This phase I trial studies the side effects and best dose of terameprocol in treating patients with high-grade glioma that has come back. Drugs used in chemotherapy, such as terameprocol, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of terameprocol given orally on days 1-5 every 28 days in patients with high grade glioma. (Part 1)

II. To evaluate terameprocol tumor to plasma ratios in resected high grade gliomas following 5 days of oral terameprocol administration. (Part 2)

III. To assess the maximum duration of terameprocol that can be safely administered on a continuous basis. (Part 3)

SECONDARY OBJECTIVES:

I. Characterize the plasma pharmacokinetic (PK) of oral terameprocol.

II. Evaluate the toxicities of oral terameprocol.

III. Assess progression-free survival.

IV. Estimate overall survival.

V. Assess tumor response.

TERTIARY OBJECTIVES:

I. Assess the contribution of cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9) genotypes on the variability of oral terameprocol pharmacokinetics.

OUTLINE: This is a dose-escalation study.

Patients receive terameprocol orally (PO) once daily (QD) on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, every 2 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed supratentorial high grade glioma (grade III or IV glioma) that is progressive or recurrent following radiation therapy and chemotherapy; patients with grade IV glioma must have progressed or recurred after initial treatment with radiation and temozolomide; patients with grade III glioma must have received at least radiation and one regimen of chemotherapy (temozolomide or procarbazine, lomustine, vincristine [PCV] regimen)

  * Patients must have measurable contrast-enhancing disease by magnetic resonance imaging (MRI) imaging within 21 days of starting treatment; patient must be able to undergo MRI of the brain with gadolinium
  * Patients may have had treatment for an unlimited number of prior relapses
  * Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

    * 12 weeks from the completion of radiation
    * 6 weeks from a nitrosourea chemotherapy
    * 3 weeks from a non-nitrosourea chemotherapy
    * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
    * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.)
    * 4 weeks from prior antiangiogenesis therapy (approved or investigational) (e.g., bevacizumab, aflibercept, ramucirumab, cediranib, cabozantinib, etc.)
  * Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
  * Patients must be 18 years of age or older
  * Absolute neutrophil count >= 1,500/mcL
  * Platelets >= 100,000/mcL
  * Hemoglobin >= 9 g/dL
  * Total bilirubin =< institutional upper limit of normal
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
  * Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
  * Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
  * Patients must be able to provide written informed consent
  * Women of childbearing potential must have a negative serum pregnancy test prior to study entry; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 30 days after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 30 days after the last dose of study drug
  * Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
  * Patients must be able to swallow oral medications
  * Part 2 (surgical) patients only: patients must be undergoing surgery that is clinically indicated as determined by their care providers; patients must be eligible for surgical resection according to the following criteria:

    * Expectation that the surgeon is able to resect at least 100 mg of tumor from enhancing tumor and at least 100 mg from non-enhancing tumor with low risk of inducing neurological injury

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Patient must not have known sensitivity to terameprocol or any formulation excipients
* Patients with (mean of triplicate) QTc(F) >/= 450mS on screening 12-lead triplicate electrocardiogram (ECG) are ineligible
* Patients must not be on any anticoagulation
* Patients on any moderate or strong cytochrome P450 family 2, subfamily C, polypeptide 9 (CYP2C9) inducer (e.g., carbamazepine, rifampin) or inhibitor (e.g., amiodarone, fluconazole) are ineligible; CYP2C9 poor metabolizers will not be excluded
* Patients on narrow-therapeutic drugs that are substrates for cytochrome P450 family 1, subfamily A, polypeptide 2 (CYP1A2), CYP2C9, cytochrome P450 family 2, subfamily C, polypeptide 19 (CYP2C19), and cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, phenytoin, pimozide, quinidine, sirolimus, tacrolimus, theophylline, tizanidine, warfarin)
* Patient must not have prior gastrointestinal (GI) surgery or GI disease that might interfere with the absorption of terameprocol
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with terameprocol
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of terameprocol (Part 1) | Day 1 - Day28 (First Cycle)
  To estimate the MTDs in terms of clinical toxicities, a modified continual reassessment method, based on that described by Piantadosi et al. will be employed. Dose escalation will be guided by observed clinical toxicity in 3 patients per dose cohort after the initial dose.
Change in terameprocol tumor to plasma concentration ratio (Part 2) | Baseline, Pre-surgery (shortly before start of surgery - within 1hr) and post surgery (as soon as practical afer completion of surgery - approx 4 hrs)
  The tumor/plasma concentration ratio will be estimated.
Maximum tolerated days of terameprocol dosing that can safely be administered on a continuous basis (Part 3) | Up to 28 days
  This is a escalation study. The escalation is the number of continuous days that terameprocol can be given. Terameprocol dose will remain constant at a fix dose everyday.

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, MD, Principal Investigator — ABTC
Locations (9):
- United States (9):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abrams Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahluwalia MS, Ozair A, Rudek M, Ye X, Holdhoff M, Lieberman FS, Piotrowski AF, Nabors B, Desai A, Lesser G, Huang RC, Glenn S, Khosla AA, Peereboom DM, Wen PY, Grossman SA. A multicenter, phase 1, Adult Brain Tumor Consortium trial of oral terameprocol for patients with recurrent high-grade glioma (GATOR). Cell Rep Med. 2024 Jul 16;5(7):101630. doi: 10.1016/j.xcrm.2024.101630. Epub 2024 Jul 1. PMID 38955178